CLINICAL TRIAL: NCT02895750
Title: Efficacity and Safety of Metformin XR in CKD Stage 1 to 3
Acronym: METXR/CKD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI2016_843_0008
Record Dates: First submitted 2016-07-26; First posted 2016-09-12 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Renal Insufficiency, Chronic
Keywords: diabetes type 2; Metformin; chronic kidney disease; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- normal to mild renal impairment (Experimental): (12 subjects): eGFR ≥ 60 (normal renal function to mild renal impairment, CKD stages 1-2) METFORMIN
  Interventions: Drug: Metformin
- mild to moderate renal impairment (Experimental): (12 subjects): eGFR 59-45 (mild to moderate renal impairment, CKD stage 3a) METFORMIN
  Interventions: Drug: Metformin
- moderate to severe renal impairment (Experimental): (12 subjects): eGFR 44-30 (moderate to severe renal impairment, CKD stage 3b) METFORMIN
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin extended release tablets (Glucophage 500 mg; 750 mg; 1,000 mg) administrated during 6 to 12 weeks (CKD1 and 3B, respectively)
  Other Names: Glucophage

SUMMARY:
There is limited data availability on effect of Metformin XR on 24-h plasma glucose, and there is no available data in chronic kidney disease (CKD). The planned study aims to provide data on glucose plasma level in relation to metformin plasma level in Diabetes Type II patients.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients aged between 18 and 80 years requiring metformin (and any other antidiabetic treatment)

Exclusion Criteria:

* Pregnancy and lactation
* Hyperlactatemia (> 2.5 mmol/L)
* No creatinine levels available since 3 months
* Severe hepatic insufficiency
* No liver function parameters available
* Need of investigation with iodized contrast media
* Hypersensitivity to metformin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2022-01-08 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of once daily Metformin XR on 24-h blood glucose control | week 12
  The blood glucose will be measured continuously throughout the study using continuous glucose monitoring (mean, range and variability in each therapeutic block).

SECONDARY OUTCOMES:
Tolerability of Metformin XR in mild to moderate (CKD) | week 0, 2, 4, 6, 8, 10 and 12
  Blood creatinine levels will be measured at the end of each therapeutic block. (week 0, 2, 4, 6, 8, 10 and 12)
Tolerability of Metformin XR in mild to moderate (CKD) 2 | week 0, 2, 4, 6, 8, 10 and 12
  blood lactate levels will be measured at the end of each therapeutic block.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Daniel LALAU, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens Picardie, Amiens, France

REFERENCES:
- [Result] Lalau JD, Bennis Y, Al-Salameh A, Hurtel-Lemaire AS, Fendri S. Pharmacodynamics and pharmacokinetics of extended-release metformin in patients with type 2 diabetes and chronic kidney disease stage 3B. Diabetes Obes Metab. 2022 Jan;24(1):166-170. doi: 10.1111/dom.14554. Epub 2021 Oct 4. No abstract available. PMID 34545662